CLINICAL TRIAL: NCT06445920
Title: Risk Factors Analysis for Clinical Important Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Gastrointestinal Surgery Based on LASSO and Stepwise Regression
Brief Title: Risk Factors Analysis for Clinical Important Postoperative Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhi-Nan Zheng, Attending doctor, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2024ZSLYEC-201
Record Dates: First submitted 2024-06-02; First posted 2024-06-06 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-06

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CIPONV: The occurrence of PONV with the simplified PONV impact scale score of 5 or more.
  Interventions: Other: No Intervention
- Non-CIPONV: There was no occurrence of PONV, or if PONV occurred, the simplified PONV impact scale score was less than 5.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Postoperative nausea and vomiting (PONV) is a distressing and common complication after surgery. The concept of clinical important PONV (CI-PONV) assesses the impact of PONV on patient-reported outcomes. This research aims to conduct an analysis of the risk factors contributing to CI-PONV utilizing the least absolute shrinkage and selection operator (LASSO) and stepwise regression techniques. All 1154 patients participating in the FDP-PONV trial are included in this study and categorized into two groups: the CI-PONV group and the non-CI-PONV group. CI-PONV is defined as the occurrence of PONV with a simplified PONV impact scale score of 5 or higher within 24 hours after surgery. The LASSO method is employed to identify the most relevant variables from an initial set of 56 related variables and stepwise regression is used to further refine the selection of the ultimate predictors.A logistic regression model was developed based on the selected factors influencing CIPONV. A nomogram was developed as a tool for clinical application.

DETAILED DESCRIPTION:
Drawing from prior studies, we conducted a sample size calculation for a predictive model using the website https://mvansmeden.shinyapps.io/BeyondEPV/. By setting the number of candidate predictors to 9, the events fraction to 0.14, and the criterion value for rMPSE to 0.04, we determined that a minimum total sample size of 900 is required, with a minimally expected event per variable of 13.9. All patients were classified into either the CI-PONV group or the non-CI-PONV group. All 56 perioperative clinical features, encompassing baseline characteristics, preoperative conditions, and intraoperative information, were considered as potential predictive factors. In the quest to uncover potential predictive factors associated with CI-PONV, we employed the least absolute shrinkage and selection operator (LASSO) to sift through clinically significant variables. Subsequently, we utilized stepwise regression based on the Akaike Information Criterion (AIC) to further refine the selection of the ultimate predictors. Finally, a logistic regression model was developed based on the selected factors influencing CIPONV. The discrimination of the model was assessed by the ROCAUC and the goodness of fit of the model was evaluated using the Hosmer-Lemeshow test and calibration plots. A nomogram based on the logistic regression model output was developed as a tool for clinical application.

ELIGIBILITY:
Inclusion Criteria:

a) age between 18 and 75 years, b) having 3 or 4 Apfel risk factors, and c) scheduled to undergo laparoscopic gastrointestinal surgical procedures under general anesthesia.

Exclusion Criteria:

a) American Society of Anesthesiologists (ASA) physical status greater than 3, b) severe hepatic dysfunction, c) contraindications to fosaprepitant, 5-HT3 receptor antagonist, or dexamethasone, d) preoperative use of medications known to have antiemetic properties, e) presence of mental disorders or inability to communicate, and f) pregnant or nursing women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 1154 patients in the FDP-PONV trial will be enrolled in this study. The FDP-PONV trial was a randomized, controlled, double-blind trial that aimed to evaluate the effectiveness and safety of fosaprepitant in managing PONV in patients undergoing laparoscopic gastrointestinal surgery. The FDP-PONV trial was approved by the Ethics Committee of the Sixth Affiliated Hospital of Sun Yat-sen University (2021ZSLYEC-78), and registered at Clinicaltrials.gov (NCT04853147).
Sampling Method: Probability Sample
Enrollment: 1154 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Clinically important postoperative nausea and vomiting (CI-PONV) | The first 24 hours after surgery
  The occurrence of PONV with the simplified PONV impact scale score of 5 or more. PONV is defined as PONV as the experience of nausea, retching, or vomiting during the first 24 hours following surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhinan Zheng, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Anesthesia, The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gan TJ, Belani KG, Bergese S, Chung F, Diemunsch P, Habib AS, Jin Z, Kovac AL, Meyer TA, Urman RD, Apfel CC, Ayad S, Beagley L, Candiotti K, Englesakis M, Hedrick TL, Kranke P, Lee S, Lipman D, Minkowitz HS, Morton J, Philip BK. Fourth Consensus Guidelines for the Management of Postoperative Nausea and Vomiting. Anesth Analg. 2020 Aug;131(2):411-448. doi: 10.1213/ANE.0000000000004833. PMID 32467512
- [Background] Eberhart LH, Mauch M, Morin AM, Wulf H, Geldner G. Impact of a multimodal anti-emetic prophylaxis on patient satisfaction in high-risk patients for postoperative nausea and vomiting. Anaesthesia. 2002 Oct;57(10):1022-7. doi: 10.1046/j.1365-2044.2002.02822.x. PMID 12358962
- [Background] Myles PS, Williams DL, Hendrata M, Anderson H, Weeks AM. Patient satisfaction after anaesthesia and surgery: results of a prospective survey of 10,811 patients. Br J Anaesth. 2000 Jan;84(1):6-10. doi: 10.1093/oxfordjournals.bja.a013383. PMID 10740539
- [Background] Shaikh SI, Nagarekha D, Hegade G, Marutheesh M. Postoperative nausea and vomiting: A simple yet complex problem. Anesth Essays Res. 2016 Sep-Dec;10(3):388-396. doi: 10.4103/0259-1162.179310. PMID 27746521
- [Background] Habib AS, Chen YT, Taguchi A, Hu XH, Gan TJ. Postoperative nausea and vomiting following inpatient surgeries in a teaching hospital: a retrospective database analysis. Curr Med Res Opin. 2006 Jun;22(6):1093-9. doi: 10.1185/030079906X104830. PMID 16846542
- [Background] Parra-Sanchez I, Abdallah R, You J, Fu AZ, Grady M, Cummings K 3rd, Apfel C, Sessler DI. A time-motion economic analysis of postoperative nausea and vomiting in ambulatory surgery. Can J Anaesth. 2012 Apr;59(4):366-75. doi: 10.1007/s12630-011-9660-x. Epub 2012 Jan 6. PMID 22223185
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Background] Zhou CM, Wang Y, Xue Q, Yang JJ, Zhu Y. Predicting early postoperative PONV using multiple machine-learning- and deep-learning-algorithms. BMC Med Res Methodol. 2023 May 31;23(1):133. doi: 10.1186/s12874-023-01955-z. PMID 37259031
- [Background] Kim JH, Cheon BR, Kim MG, Hwang SM, Lim SY, Lee JJ, Kwon YS. Postoperative Nausea and Vomiting Prediction: Machine Learning Insights from a Comprehensive Analysis of Perioperative Data. Bioengineering (Basel). 2023 Oct 1;10(10):1152. doi: 10.3390/bioengineering10101152. PMID 37892882
- [Background] Edgman-Levitan S, Schoenbaum SC. Patient-centered care: achieving higher quality by designing care through the patient's eyes. Isr J Health Policy Res. 2021 Mar 5;10(1):21. doi: 10.1186/s13584-021-00459-9. PMID 33673875
- [Background] Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth. 2012 Mar;108(3):423-9. doi: 10.1093/bja/aer505. Epub 2012 Jan 29. PMID 22290456
- [Background] Hubbard RA, Su YR, Bowles EJA, Ichikawa L, Kerlikowske K, Lowry KP, Miglioretti DL, Tosteson ANA, Wernli KJ, Lee JM. Predicting five-year interval second breast cancer risk in women with prior breast cancer. J Natl Cancer Inst. 2024 Jun 7;116(6):929-937. doi: 10.1093/jnci/djae063. PMID 38466940
- [Background] Liu J, Yu Y, Qi W, Ma X, Han Y. Innovation and entrepreneurship of Chinese returning migrant workers in their home region. Heliyon. 2024 Apr 26;10(9):e30296. doi: 10.1016/j.heliyon.2024.e30296. eCollection 2024 May 15. PMID 38694132
- [Background] Portet S. A primer on model selection using the Akaike Information Criterion. Infect Dis Model. 2020 Jan 7;5:111-128. doi: 10.1016/j.idm.2019.12.010. eCollection 2020. PMID 31956740